CLINICAL TRIAL: NCT02266875
Title: Nebulized Hypertonic Saline for Inpatient Use in Chronic Obstructive Pulmonary Disease
Brief Title: Nebulized Hypertonic Saline for Inpatient Use in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0050
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic Saline (Experimental): Patients will receive nebulized hypertonic (3%) saline along with standard 2.5 mg. albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
  Interventions: Drug: hypertonic saline
- Standard Saline (Active Comparator): Patients will receive standard saline (0.9%) saline along with standard 2.5 mg. albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
  Interventions: Drug: standard saline

INTERVENTIONS:
Drug: hypertonic saline
  Arms: Hypertonic Saline
Drug: standard saline
  Arms: Standard Saline

SUMMARY:
A comparison of albuterol treatments using hypertonic saline (3%) versus standard saline (0.9%) in patients with admitted patients COPD in regard to Modified Borg Dyspnea scale scores after 4 treatments within 24 hours.

DETAILED DESCRIPTION:
Hypothesis:

A clinically significant difference exists between albuterol treatments with nebulized 3% saline versus standard saline, for improvements in the patient's modified Borg dyspnea score during an acute exacerbation of COPD.Study

Population:

This study will involve 146 patients admitted to Doctors Hospital in Columbus, Ohio from September 2014 through September 2015 with a clinical diagnosis of an acute exacerbation of COPD, defined as an increase in the patient's dyspnea, cough, or change in sputum consistency/volume/color from the patient's baseline during stable conditions.

Study Design:

Patients will be randomly assigned to 2.5 mg albuterol treatments with either normal saline, as is the standard, or hypertonic saline.

Once the patient is enrolled, they will be randomly assigned to 2.5 mg albuterol treatments with either normal saline, as is the standard, or hypertonic saline. They will then receive the 2.5mg albuterol treatment, and saline solution as determined by the randomization plan (Group 1 will receive 0.9% saline and Group 2 will receive 3% saline), every six hours for at least the first 24 hours, with allowance for PRN (pro re nata= as needed) use every four hours by patient request.

The patient's dyspnea will be evaluated prior to starting the treatment and after the intervention period is completed using the Modified Borg Dyspnea Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Admitted to Doctors Hospital with a clinical diagnosis of COPD
* Documented obstruction on spirometry from prior records available at the time of the study.

Exclusion Criteria:

* Patients younger than 18 years of age
* Spirometry data not available
* History of smoking less than twenty pack-years
* Possibility of other primary cause of the patient's change in dyspnea or cough (e.g. pneumonia, congestive heart failure with pulmonary edema, myocardial infarction)
* Patient is found to have a different primary cause after initial enrollment
* Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kruti Patel, DO, Principal Investigator — OhioHealth
Locations (1):
- Doctors Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic Saline: Patients will receive nebulized hypertonic (3%) saline along with standard 2.5 mg. albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
  hypertonic saline
- Standard Saline: Patients will receive standard saline (0.9%) saline along with standard 2.5 mg. albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
  standard saline
Period: Overall Study
Arm/Group | Hypertonic Saline | Standard Saline
Started | 40 | 30
Completed | 29 | 30
Not Completed | 11 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | Standard Saline | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (8.4) | 63.3 (9.8) | 61.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 16 | 13 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-treatment Score: Modified Borg Dyspnea Scale [Mean (Standard Deviation); unit: units on a scale] — This is a patient-reported scale to rate the difficulty of breathing. The scale ranges from 0 to 10, wherein "0" indicates no difficulty breathing, and "10" indicates a maximal difficulty in breathing.
  Patients may report in whole numbers, from 0 to 10, in addition to reporting 0.5, which indicates "very, very slight (just noticeable) difficulty in breathing."
  units on a scale | 5.1 (1.6) | 4.4 (2.2) | 4.8 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Breathing Difficulty - Using Modified Borg Dyspnea Scale
Description: This is a patient-reported scale to rate the difficulty of breathing. The scale ranges from 0 to 10, wherein "0" indicates no difficulty breathing, and "10" indicates a maximal difficulty in breathing. Patients may report in whole numbers, from 0 to 10, in addition to reporting 0.5, which indicates "very, very slight (just noticeable) difficulty in breathing."
  A negative change in score indicates a reduction in patient-reported breathing difficulty. The greater the negative change, the better the patient-reported breathing.
Time Frame: Pre-treatment (baseline) vs. 24 hours post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypertonic Saline | Standard Saline
Number analyzed (Participants) | 29 | 30
units on a scale | -1.4 (1.6) | -1.0 (2.1)
Statistical Analysis 1: Comparison: Hypertonic Saline vs Standard Saline; Test type: Superiority; p = 0.320, t-test, 2 sided

2. Secondary Outcome: 30 Day Readmission
Description: Documented hospital readmission 30 days post discharge
Time Frame: 30 days post discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | Standard Saline
Number analyzed (Participants) | 29 | 30
Participants | 3 | 3
Statistical Analysis 1: Comparison: Hypertonic Saline vs Standard Saline; Test type: Superiority; p > 0.999, Fisher Exact

3. Secondary Outcome: 30 Day All Cause Mortality
Description: Documented mortality at 30 days post discharge
Time Frame: 30 days post discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | Standard Saline
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected during subject admission period, from the time of study enrollment (baseline) until they were discharged from the hospital, ending their study participation.
Groups:
- Hypertonic Saline: Patients will receive nebulized hypertonic (3%) saline along with standard 2.5 mg albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
- Standard Saline: Patients will receive standard saline (0.9%) saline along with standard 2.5 mg albuterol treatments once every 6 hours for 24 hour, with allowance for PRN (as needed use).
  Dyspnea will be assessed prior to treatment and at completion of the 24 hour period using the Modified Borg Dyspnea Scale.
Arm/Group | Hypertonic Saline | Standard Saline
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT02266875/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT02266875/ICF_001.pdf